CLINICAL TRIAL: NCT06650995
Title: AlEX-DHF: Ablation and Exercise in Diastolic Heart Failure
Acronym: AlEX-DHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-381-S-SB
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction; Atrial Fibrillation
Keywords: exercise capacity; ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1:1 randomization will be done into interventional and control groups with the aid of sealed envelopes
Who Masked: Investigator
Masking Description: The principal investigator (PI) will not receive information on group allocation. Group allocation and data will be saved in a password-secured database, which will not be accessible to the PI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group receives exercise training
  Interventions: Other: Exercise training
- Control Group (No Intervention): This group does not receive exercise training

INTERVENTIONS:
Other: Exercise training — exercise intervention will consist of supervised, home-based, combined training with elements of endurance, resistance and respiratory training
  Arms: Intervention Group

SUMMARY:
The investigators analyze the impact of exercise and ablation in patients with symptomatic short-persistent atrial fibrillation (Afib) and heart failure with preserved ejection fraction (HFpEF). It is hypothesized that the combination of ablation and exercise better improves peak oxygen consumption (VO2peak) through improvement of peripheral (exercise training) and central (ablation) adaptations.

Exercise intervention will contain a 12-week combined, video-based, supervised, endurance, resistance and respiratory training.

DETAILED DESCRIPTION:
In a feasibility study the investigators analyze the impact of exercise and ablation in patients with symptomatic short-persistent atrial fibrillation and heart failure with preserved ejection fraction. Patients will be randomized into 2 groups: (1) A control group receiving ablation therapy, and (2) a group receiving ablation therapy and a combination of endurance, strength and respiratory training. The investigators will include 20 patients/group. All patients will receive a smart watch to monitor heart rate and trigger ECG recordings during symptomatic episodes. Smart watch monitoring will be done for 4 weeks. Then all patients will receive baseline examination with laboratory markers, lung function testing, echocardiography, measurement of pulse wave velocity, and screening for sleep apnea. All patients will receive simultaneous cardiopulmonary exercise testing (CPET) and exercise right heart catheterization (exRHC) followed by ablation therapy. Patients will then be randomized into a training and control group. After 2 weeks all patients will receive outpatient CPET to assess changes of VO2peak compared to baseline.

The training group will receive home-based, video-supervised exercise training with a combination of endurance, strength and respiratory training (5x/week). The control group will receive standard recommendations on physical activity. Smart watch monitoring will be continued in all groups until the end of the study. After 12 weeks of training intervention, all groups will undergo echocardiography, lung function testing, measurement of pulse wave velocity and exRHC with simultaneous CPET. All patients will receive 24h Holter monitoring at the end of the study. During exRHC lactate kinetics will be analyzed and improvement of lactate thresholds through exercise training will be determined. The primary outcome is the improvement of VO2peak in the groups. Secondary outcomes are improvements in the ratio of pulmonary capillary wedge pressure/cardiac output (PAWP/CO) and mean pulmonary artery pressure/CO (mPAP/CO). Burden of atrial fibrillation in the groups will also be assessed. All groups will receive optimal drug therapy.

The investigators expect that a combined approach of ablation and exercise training will better improve VO2peak through central (ablation) and peripheral (exercise training) adaptations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed heart failure with preserved ejection fraction
* Symptomatic short-persistent atrial fibrillation (diagnosis within 1 year of study inclusion)

Exclusion Criteria:

* Paroxysmal, long-persistent or permanent atrial fibrillation
* Clinically unstable coronary artery disease or acute coronary syndrome
* Physical and/or mental inability to perform exercise testing
* Prior ablation therapy
* Precapillary pulmonary hypertension at rest
* Intracardiac shunts
* Left ventricular ejection fraction <50%
* High-degree valve insufficiency or stenosis (greater than grade 1 at rest)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Delta of peak oxygen consumption | 14 weeks
  Improvement of peak oxygen consumption between baseline and after 12 weeks of training

SECONDARY OUTCOMES:
Delta of mean pulmonary artery pressure and cardiac output (mPAP/CO) | 14 weeks
  Improvement of delta mPAP/CO between baseline and after 12 weeks of training
Delta of pulmonary artery wedge pressure to cardiac output (PAWP/CO) | 14 weeks
  Improvement of delta PAWP/CO between baseline and after 12 weeks of training
Delta of peak oxygen consumption baseline to post ablation | 2 weeks
  Improvement of peak oxygen consumption from baseline to post ablation
Delta of peak oxygen consumption post ablation to the end of the study | 12 weeks
  Improvement of peak oxygen consumption from post ablation to the end of the study
Delta of Kansas City Cardiomyopathy Questionnaire score | 14 weeks
  Difference in the score between baseline and after 12 weeks of training (values ranging from 0-100; a higher score being associated with better quality of life in patients with heart failure)
Delta of E/e' | 14 weeks
  Difference of E/e' between baseline and after 12 weeks of training
Burden of atrial fibrillation in the groups | 18 weeks
  Difference of episodes of atrial fibrillation between the groups. Episodes of atrial fibrillation will be counted numerically with telemetry. Patients will trigger ECG recordings with their smart watch at three time points a day (8am, 2pm, 8pm) regardless of symptoms, and whenever symptoms occur (palpitations, dizziness, dyspnea, chest discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Wernhart, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Department of Medicine, Division of Prevention and Sports Medicine TU Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No
Information can be received on reasonable request from the principal investigator

REFERENCES:
- [Result] Wernhart S, Goertz A, Hedderich J, Papathanasiou M, Hoffmann J, Rassaf T, Luedike P. Diastolic exercise stress testing in heart failure with preserved ejection fraction: The DEST-HF study. Eur J Heart Fail. 2023 Oct;25(10):1768-1780. doi: 10.1002/ejhf.2995. Epub 2023 Aug 24. PMID 37565370
- [Result] Anker SD, Usman MS, Anker MS, Butler J, Bohm M, Abraham WT, Adamo M, Chopra VK, Cicoira M, Cosentino F, Filippatos G, Jankowska EA, Lund LH, Moura B, Mullens W, Pieske B, Ponikowski P, Gonzalez-Juanatey JR, Rakisheva A, Savarese G, Seferovic P, Teerlink JR, Tschope C, Volterrani M, von Haehling S, Zhang J, Zhang Y, Bauersachs J, Landmesser U, Zieroth S, Tsioufis K, Bayes-Genis A, Chioncel O, Andreotti F, Agabiti-Rosei E, Merino JL, Metra M, Coats AJS, Rosano GMC. Patient phenotype profiling in heart failure with preserved ejection fraction to guide therapeutic decision making. A scientific statement of the Heart Failure Association, the European Heart Rhythm Association of the European Society of Cardiology, and the European Society of Hypertension. Eur J Heart Fail. 2023 Jul;25(7):936-955. doi: 10.1002/ejhf.2894. Epub 2023 Jul 17. PMID 37461163
- [Result] Houstis NE, Eisman AS, Pappagianopoulos PP, Wooster L, Bailey CS, Wagner PD, Lewis GD. Exercise Intolerance in Heart Failure With Preserved Ejection Fraction: Diagnosing and Ranking Its Causes Using Personalized O2 Pathway Analysis. Circulation. 2018 Jan 9;137(2):148-161. doi: 10.1161/CIRCULATIONAHA.117.029058. Epub 2017 Oct 9. PMID 28993402
- [Result] Jain CC, Borlaug BA. Hemodynamic assessment in heart failure. Catheter Cardiovasc Interv. 2020 Feb 15;95(3):420-428. doi: 10.1002/ccd.28490. Epub 2019 Sep 10. PMID 31507065
- [Result] Mueller S, Winzer EB, Duvinage A, Gevaert AB, Edelmann F, Haller B, Pieske-Kraigher E, Beckers P, Bobenko A, Hommel J, Van de Heyning CM, Esefeld K, von Korn P, Christle JW, Haykowsky MJ, Linke A, Wisloff U, Adams V, Pieske B, van Craenenbroeck EM, Halle M; OptimEx-Clin Study Group. Effect of High-Intensity Interval Training, Moderate Continuous Training, or Guideline-Based Physical Activity Advice on Peak Oxygen Consumption in Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2021 Feb 9;325(6):542-551. doi: 10.1001/jama.2020.26812. PMID 33560320
- [Result] Rattka M, Pott A, Kuhberger A, Weinmann K, Scharnbeck D, Stephan T, Baumhardt M, Bothner C, Iturbe Orbe M, Rottbauer W, Dahme T. Restoration of sinus rhythm by pulmonary vein isolation improves heart failure with preserved ejection fraction in atrial fibrillation patients. Europace. 2020 Sep 1;22(9):1328-1336. doi: 10.1093/europace/euaa101. PMID 32449907
- [Result] Rattka M, Kuhberger A, Pott A, Stephan T, Weinmann K, Baumhardt M, Aktolga D, Teumer Y, Bothner C, Scharnbeck D, Rottbauer W, Dahme T. Catheter ablation for atrial fibrillation in HFpEF patients-A propensity-score-matched analysis. J Cardiovasc Electrophysiol. 2021 Sep;32(9):2357-2367. doi: 10.1111/jce.15200. Epub 2021 Aug 18. PMID 34379370
- [Result] Wernhart S, Papathanasiou M, Mahabadi AA, Rassaf T, Luedike P. Betablockers reduce oxygen pulse increase and performance in heart failure patients with preserved ejection fraction. Int J Cardiol. 2023 Jan 1;370:309-318. doi: 10.1016/j.ijcard.2022.10.009. Epub 2022 Oct 8. PMID 36220507
- [Result] Wernhart S, Oster M, Schulze M, Papathanasiou M, Ruhparwar A, Rassaf T, Luedike P. Moderate Continuous and Modified High-Intensity Interval Training in Patients With Left Ventricular Assist Devices: The Prospective Train-the-LVAD Trial. J Card Fail. 2023 May;29(5):841-848. doi: 10.1016/j.cardfail.2023.01.007. Epub 2023 Feb 8. PMID 36758740